CLINICAL TRIAL: NCT03985202
Title: Can a Structured Exercise Programme Improve the Predicted Survival for Planned Abdominal Aortic Aneurysm Surgery Patients?
Brief Title: Structured Exercise Programme and Abdominal Aortic Aneurysm Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS194690
Record Dates: First submitted 2019-06-04; First posted 2019-06-13 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: exercise programme
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Non-randomised interventional observational study. Pilot study. 60 patients to be recruited from the Torbay AAA screening programme and AAA surveillance group over a two-year period.
  Cardiopulmonary exercise test and survival prediction when AAA reaches 4.5 cm. (Current clinical practice).
  9 week structured exercise programme. 3 sessions per week. (Intervention). Repeat cardiopulmonary exercise test and survival prediction after structured exercise programme. Advice given for on going exercise and maintenance of fitness. (Intervention).
  Repeat cardiopulmonary exercise test and survival prediction after 3 months after structured exercise programme. (Intervention).
  Pateitns are asked to complete the following questionnaires:- EQ-5D-5L and Hospital Anxiety and Depression Scale (HADS) before, after the last exercise session and 3 months after the exercise programme. Change in medical or drug history. Change in weight or smoking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Structured Exercise Programme (Experimental): An initial 45 min exercise counselling incorporating behaviour modification techniques.
  Participants will be offered three sessions per week of aerobic interval exercise on a cycle ergometer over nine weeks. Exercise programmes will be tailored to each patient, taking previous level of activity, mobility and any barriers to exercise into consideration.
  Following this:
  Participants will be encouraged to comply with current physical activity recommendations: 150 min of moderate intensity aerobic exercise per week (brisk walking / cycling). They will also be sign posted to local exercise facilities.
  Interventions: Other: Structured exercise programme

INTERVENTIONS:
Other: Structured exercise programme — 9 week structured exercise programme. 3 sessions per week. (Intervention).The patient will be invited to the hospital for a 45-minute exercise counselling session, incorporating behaviour modification techniques. These behaviour modification techniques will be reinforced during the supervised exercise sessions. Participants will be offered 3 sessions of supervised aerobic interval exercise sessions per week on a cycle ergometer for 9 weeks.Exercise programmes will be tailored to each patient, taking previous level of activity, mobility and any barriers to exercise into consideration.
  Other Names: Qualitiative interviews and questionnaires

SUMMARY:
There is a relationship between aerobic fitness and survival both with and without surgery. Some patients can improve their aerobic fitness with a structured exercise programme but currently it is not know how much this could change predicted survival for patients with an abdominal aortic aneurysm, or how long this change can be maintained. Survival can be predicted after planned abdominal aortic aneurysm (AAA) surgery using physical fitness measured with a cardiopulmonary exercise test. The researchers have validated this in a published peer reviewed multicentre study. In this study the patient's fitness will be measured before and after a structured exercise programme and assess if there is any change in their predicted survival. The primary objective of the study is to measure the change in predicted survival for abdominal aortic aneurysm surgery after a structured exercise programme. In addition the patients are asked to complete the following questionnaires:- EQ-5D-5L, Hospital Anxiety and Depression Scale (HADS) before and after the exercise programme.

DETAILED DESCRIPTION:
The UK has a national AAA screening programme. At the age of 65 men are offered a one off ultrasound test to look for a AAA. If their abdominal aorta is > 5.5 cm they are referred to a Vascular Surgeon. If the patients abdominal aorta is between 3 cm and 5.4 cm they are offered further ultrasound scans to monitor the size of their aorta. This is a surveillance programme. In addition men who have an AAA between 3 cm and 5.4 cm that is detected by an ultrasound scan, CT or MRI performed as part of an investigation for another clinical problem are added to the surveillance programme.

In Torbay and South Devon men in the AAA surveillance programme are referred for a Cardiopulmonary Exercise Test when the AAA reaches 4.5 cm as part of standard clinical practice. This takes place in the Pre assessment Clinic in Torbay Hospital and is performed by a Consultant Anaesthetist. If the patient is able to safely perform the Cardiopulmonary Exercise Test they will be identified as potential participants by the Consultant Anaesthetist.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants ≥ 18
2. Under surveillance as part of the AAA screening or surveillance programme with an AAA that is between 4.5 cm and 5.4 cm
3. Able and willing to provide informed consent
4. Understand verbal and written instructions in English
5. Able to safely perform a cardiopulmonary exercise test (this will confirm they can use a cycle ergometer)
6. Patients who are already participating (or have participated) in other trials may be eligible, but the relevant trial teams must agree this in advance.-

Exclusion Criteria:

1. Contra-indications to exercise (lower limb amputation without prosthesis, bone, joint or muscle problem which may be exacerbated by exercise, chronic lung disease causing desaturation with exercise or shortness of breath at rest, severe psychiatric health problems)
2. Cardiovascular contra-indications (unstable angina, acute left ventricular failure, uncontrolled cardiac arrhythmias, uncontrolled hypertension, cardiac event in the previous 6 weeks, cerebral vascular accident in the previous 6 weeks)
3. Participation in other treatment trials, where this has not been agreed in advance with both trial teams
4. Symptomatic AAA
5. Urgency of surgery for AAA precludes undertaking exercise programme. -

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in predicted mortality: 30- day postoperative mortality (%) or median survival (years). | 3 months post end of exercise programme
  We can predict survival after planned abdominal aortic aneurysm (AAA) surgery using physical fitness measured with a cardiopulmonary exercise test, age and comorbidities. We have validated this in a published peer reviewed multicentre study. We will measure patient's fitness before and after a structured exercise programme and assess if there is any change in their predicted survival. The primary objective of the study is to measure the change in predicted survival for abdominal aortic aneurysm surgery after a structured exercise programme.

SECONDARY OUTCOMES:
Change in Health related Quality of Life (HRQoL) scores | 1 week and 3 months post end of exercise programme
  Metric: Completion of EuroQol EQ5D-5L questionnaires before the structured exercise programme, within a week of the end of the exercise programme and 3 months after the end of the exercise programme
Change in Psychological Health Status | 1 week and 3 months post end of exercise programme
  Metric: Completion of Hospital Anxiety and Depression (HAD) questionnaire before the structured exercise programme, within a week of the end of the exercise programme and 3 months after the end of the exercise programme
Change in weight | 1 week and 3 months post end of exercise programme
  Metric: Change in weight before the structured exercise programme, within a week of the end of the exercise programme and 3 months after the end of the exercise programme
Change in cardiopulmonary exercise test | 1 week and 3 months post end of exercise programme
  Metric: Change in cardiopulmonary fitness variables (VO2, anearobic threshold, VE/VCO2,oxygen pulse), as measured using an incremental Cardiopulmonary exercise test (CPET) before the structured exercise programme, within a week of the end of the exercise programme and 3 months after the end of the exercise programme
Change in smoking status | 1 week and 3 months post end of exercise programme
  Metric: Change in smoking habits (stopped, reduced) before the structured exercise programme, within a week of the end of the exercise programme and 3 months after the end of the exercise programme

CONTACTS AND LOCATIONS:
Locations (1):
- Torbay Hospital, Torquay, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No